CLINICAL TRIAL: NCT02324400
Title: Pilot Study for the Evaluation of the Safety and Performance of the RenaSense System in Hospitalized Acute Decompensated Heart Failure Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nephera Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRNS003
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Heart Decompensation; Heart Failure, Congestive; Renal Insufficiency
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator)
  Interventions: Device: RenaSense Stimulation
- Control (Sham Comparator)
  Interventions: Device: RenaSense Sham Control

INTERVENTIONS:
Device: RenaSense Stimulation — RenaSense Catheter, Electrical Stimulation of the Urinary Bladder Wall
  Arms: Treatment
Device: RenaSense Sham Control — RenaSense Catheter,no delivery of stimulation
  Arms: Control

SUMMARY:
The study is intended to verify the safety and assess the performance of up to 3-days treatment protocol with the RenaSense System in ADHF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Females
2. Age 18-85 years
3. Admitted to the hospital with a primary diagnosis of decompensated heart failure
4. Estimated glomerular filtration rate (GFR)* ≤60 ml/min and ≥20 ml/min, based on serum creatinine at initial evaluation
5. History of chronic use of oral loop diuretics (≥ 80 mg/day Furosemide or equivalent) during the past 3 months
6. Indication for treatment with intravenous diuretics
7. Volume overload

   For patients with a pulmonary artery catheter, persistent volume overload will include:
   * Pulmonary capillary wedge pressure greater than 22mmHg and one of the following clinical signs:
   * at least 2+ peripheral edema and/or
   * Pulmonary edema or pleural effusions on chest x-ray

   For patients without a pulmonary artery catheter, persistent volume overload will include at least two of the following:
   * At least 2+ peripheral edema
   * Jugular venous pressure greater than 10 cm on physical examination (or central venous pressure greater than 10 mmHg when measured)
   * pulmonary edema or pleural effusions on chest x-ray
8. Indication for urinary catheterization
9. BNP > 400 pg/mL at initial evaluation
10. Able and willing to sign the informed consent

Exclusion Criteria:

1. History of urinary tract infection within the last 1 month based on medical history and/or urinalysis on day of admission
2. Gross hematuria, perineal hematoma or symptomatic microscopic hematuria
3. Hypertension, systolic >180 mmHg or diastolic > 110 mmHg
4. Hypotension, systolic pressure <100 mmHg
5. Status post renal denervation
6. Implanted cardiac rhythm management device such as pacemakers, cardiac resynchronization therapy (CRT), Implantable cardioverter-defibrillator (ICD)
7. Suspected or known pregnancy
8. Previous organ transplantation
9. Life threatening condition such as severe infection, malignancy or infarction
10. Subject is participating in other concurrent clinical investigation
11. Diseases or conditions which, in the judgment of the investigator, preclude participation in the clinical trial

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with unanticipated adverse events as a measure of safety and tolerability | 72 hours

SECONDARY OUTCOMES:
Renal Function as Assessed by Serum Cystatin C level | 24, 48 and 72 hours
Urinary symptoms, hospitalizations and mortality | 90 days
  Assess no increase in urinary symptoms of obstruction or incontinence, hospitalizations and mortality rates following 30 days and 90 days follow-up, as compared to control with no electrical stimulation treatment
Sum of Global Rank Score following 72 hours of treatment as compared to baseline | 72 hours
Urine volume | 24, 48 and 72 hours
  Urine output volume collected over 24 hour intervals during days 1 to 3 of treatment

OTHER OUTCOMES:
Dosage of Furosemide administration | 72 hours
Dyspnea score as assessed by Likert scale | 72 hours
Body weight | 72 hours
Fractional excretion of Sodium | 24, 48 and 72 hours
Serum brain natriuretic peptide (BNP) values following 48 and 72 hours of treatment | 48 and 72 hours
Urine Neutrophil Gelatinase-Associated Lipocalin (NGAL) following 72 hours of treatment as compared to baseline | 72 hours

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Rambam Health Care Campus, Haifa, Outside USA
  - Hillel Yaffe Medical Center, Hedera
  - Ziv Medical Center, Safed